CLINICAL TRIAL: NCT00774449
Title: Characterization of Bronchiolitis-obliterans Syndrome (BOS) Following Lung Transplantation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hannover Medical School (Other)
Responsible Party: Dr. Jens Gottlieb, Hannover Medical School, Department of Respiratory Medicine
Other Study IDs: 5108
Record Dates: First submitted 2008-10-16; First posted 2008-10-17 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2009-07

CONDITIONS: Lung Transplantation; Bronchiolitis Obliterans Syndrome
Keywords: lung transplantation; bronchiolitis obliterans syndrome; broncholaveolar lavage; high-resolution computertomography; quality of life
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — bronchoalveolar lavage, transbronchial biopsies, blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: individuals, who have undergone double (DLTx) or heart and lung transplantation (HLTx) at Hannover Medical School 6 months prior to inclusion

SUMMARY:
Chronic organ dysfunction after lung transplantation (BOS) is the most common cause of death in long-term survivors after lung transplantation and refractory to most interventions. Early markers will be established in this project study to overcome the problem of disease recognition when impairment of graft function is already taken place. Long-term longitudinal monitoring in stable recipients of innovative markers of airway inflammation and ventilation and new imaging techniques will define different entities of chronic organ dysfunction after LTx. A database and specimen service unit for further projects will be created.

Hypothesis: This project will reveal new markers and imaging tools in recipients who develop BOS after lung transplantation. These tools will allow earlier diagnosis and more accurate monitoring of the disease process. Different patterns of the disease will be characterized.

DETAILED DESCRIPTION:
Chronic organ dysfunction of the lung allograft is the most common cause of death in lung transplant recipients after the first postoperative year and is a major cause of morbidity in the long-term care. It affects every second recipient surviving 5 years after transplantation (Boehler, Estenne 2003). Obliterative bronchiolitis (OB) is the histo-pathological process underlying chronic organ dysfunction after LTx. Bronchiolitis obliterans syndrome (BOS) is the clinical definition of chronic organ dysfunction following lung transplantation (LTx) and refers to a progressive obstructive ventilatory disorder. Staging is performed according to baseline values of forced expiratory volume after LTx (Estenne et al. 2001).

Excessive immunosuppression may be deleterious by increasing the risk of infection, thereby triggering innate and adaptive immunity. BOS is progressive in most of the cases with stabilisation in some. Different clinical entities are found according to time of onset, speed of decline in graft function (Jackson et al. 2002), ventilatory patterns, findings on imaging studies (Pakhale et al 2005, Choi et al 2003) and response to macrolides (Gerhardt et al. 2003). Exhaled biomarkers are promising markers of disease activity in pats with BOS (an Muylem 2007, Brugiere et al 2005) Alloimmune-independent and -dependent mechanisms produce injuries and inflammation of epithelial cells and subepithelial structures, leading to aberrant tissue repair (Nicod et al 2006). The triggering of innate immunity by various infections (especially respiratory viruses, Khalifah et al 2004) or chemical injuries (e.g. gastroesophageal reflux or aspiration, Palmer et al. 2000), may lead to the release of danger signals that are able to activate dendritic cells, a crucial link with adaptive immunity. Inflammation can also increase the expression and display of major histocompatibility alloantigens and thus favor the initiation of rejection episodes. The injuries evoke a proinflammatory response and cellular infiltration that leads to excessive fibroproliferation and results in matrix deposition and vascular remodelling. These phenomena may be limited in time and location or may be protracted. Reducing the risk of alloimmune-independent factors may be as important as treating acute episodes of lung rejection.

Newpotential therapeutic targets are emerging from the research performed on leukotriene receptors, chemokine receptors, and growth factors. Neutralizing these molecules may reduce the initial mononuclear and polynuclear infiltrates or the subsequent fibroproliferative process and the neovascular changes, feeding this process. (Nicod 2006). Macrolides are promising new agents which partially reverse loss of graft function in a subgroup of patients, which may change definition of BOS in the near future (Gerhardt et al 2003).

ELIGIBILITY:
Inclusion Criteria:

* Individuals, who have undergone double (DLTx) or heart and lung transplantation (HLTx) at Hannover Medical School 6 months prior to inclusion
* Ages: 18 to 68 Years
* Gender: both
* Stable graft function (FEV1 >90% baseline)

Exclusion Criteria:

* Severe airway complications after surgery necessitating repeated intervention during the last 3 months
* Need for supplemental oxygen at time of inclusion
* Single lung (SLTx) and living lobar recipients
* Established diagnosis of BOS at time of inclusion
* Inability to undergo bodyphlethysmography e.g. due to persistent infection with multi-drug resistant bacteria (MRSA, VRE, Burkholderia Cepacia, Pandorea)

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: individuals, who have undergone double (DLTx) or heart and lung transplantation (HLTx) at Hannover Medical School 6 months prior to inclusion
Sampling Method: Non-Probability Sample
Enrollment: 261 (Estimated)
Dates: Start 2009-07; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Bronchiolitis obliterans Syndrom (BOS) | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jens Gottlieb, MD, Principal Investigator — Hannover Medical School
Locations (1):
- Department of Respiratory Medicine, Medizinische Hochschule Hannover, Hanover, Germany